CLINICAL TRIAL: NCT04416919
Title: A Proposed Alternative to the N-95 Mask Shortage in the COVID-19 Pandemic. A Feasibility Study
Brief Title: Assessment of N-95 Facemask for Use in COVID-19 Pandemic in Case of Shortage of Personal Protective Equipment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 11887
Record Dates: First submitted 2020-05-13; First posted 2020-06-04 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Coronavirus Infection; Disease Prevention
Keywords: 2019 novel coronavirus disease; 2019 novel coronavirus infection; COVID-19 pandemic; COVID-19 virus disease; COVID19; COVID-19 virus infection; N-95; Respiratory protective devices; Protection from respiratory infecton; Safety; Efficacy; Pandemic
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assembled Mask (Other): Participant will be fitted with a full-face mask that covers the mouth and nose or a Whole face mask that covers the eyes, nose, and mouth depending on participant's preferences. The Fitted Mask will be attached to a bacterial/viral filter for fit testing. After completing the Fit test, the mask will be placed on the face for 15 minutes while the participant performs various activities to document the ability to tolerate the respirator. Participants oxygen and carbon dioxide level will be measured in the beginning and at the end of the 15 minutes. The individuals will be able to remove the Mask anytime if they experience significant discomfort or claustrophobia. At the end, the mask will be removed.
  Interventions: Other: Assembled mask

INTERVENTIONS:
Other: Assembled mask — Assembled masks consisting of 3 parts: A facemask (Respironics Performax Whole Face Mask or Hans Rudolph mask naso-oral mask) linked by a blue elbow ( RP Performax SE ELBOW) to a ventilator filter (Teleflex Bacterial/Viral filter 1605 or Iso-Gard HEPA light Filter 28022)

SUMMARY:
The purpose of this study is to assess the safety and efficiency of an assembled modified mask in protecting health care workers against Coronavirus in case of any personal protective equipment shortage. At least 20 healthy participants will be recruited to try the modified mask. The modified masks will be made from masks that are already available as well as filters available in the pulmonary department at the Oklahoma City VA Health Care System

ELIGIBILITY:
Inclusion Criteria:

1. All individuals older than 18 years of age, and willing to participate in the study

Exclusion Criteria:

1. Individuals with known severe COPD/emphysema, Obesity Hypoventilation or hypercapnic condition
2. Individuals with allergy or reactions to latex or masks
3. Individuals reporting dyspnea or unable to breathe comfortably in these masks
4. Claustrophobic individuals
5. Inability to create a proper Seal while inhaling through a closed filter (See Below)
6. Individuals who cannot safely apply and remove these masks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Success Percentage | 15 minutes
  Conduct a quantitative fit test and calculate the percentage of participants who pass the test.

SECONDARY OUTCOMES:
End-tidal CO2 Variation. Description: mmHg. | at 0 and 15 minutes
  Change in end-tidal CO2 from 0 to 15 minutes while wearing the Full or the Whole mask
Oxygen Pulse Oximetry Variation. Description: mmHg. | at 0 and 15 minutes.
  Measure the change in Oxygen Pulse Oximetry from 0 to15 minutes while wearing the Full or the Whole mask
Mask Visibility. Description: Likert Scale. | 15 minutes
  Evaluate the visibility (5-point Likert scale from Absent to Complete) while wearing the Full or the Whole mask for 15 minutes
Willingness of usage. Description: Likert Scale. | after 15 minutes
  When the mask is removed, participants will be asked about willingness to use this mask compared to N-95 masks using a 5-point Likert scale from 'Very unlikely' to 'Very likely'.

CONTACTS AND LOCATIONS:
Overall Officials: Houssein Youness, MD, Principal Investigator — University of Oklahoma HSC - OKC Veterans Affairs Medical Center
Locations (1):
- Oklahoma City VA Health Care System, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prevention CfDCa. Strategies for Optimizing the Supply of Facemasks: COVID-19. https://www.cdc.gov/coronavirus/2019-ncov/hcp/ppe-strategy/face-masks.html
- [Result] van Doremalen N, Bushmaker T, Morris DH, Holbrook MG, Gamble A, Williamson BN, Tamin A, Harcourt JL, Thornburg NJ, Gerber SI, Lloyd-Smith JO, de Wit E, Munster VJ. Aerosol and Surface Stability of SARS-CoV-2 as Compared with SARS-CoV-1. N Engl J Med. 2020 Apr 16;382(16):1564-1567. doi: 10.1056/NEJMc2004973. Epub 2020 Mar 17. No abstract available. PMID 32182409
- [Result] Qian Y, Willeke K, Grinshpun SA, Donnelly J, Coffey CC. Performance of N95 respirators: filtration efficiency for airborne microbial and inert particles. Am Ind Hyg Assoc J. 1998 Feb;59(2):128-32. doi: 10.1080/15428119891010389. PMID 9487666